CLINICAL TRIAL: NCT07297147
Title: Do Dental Implants Move During Osseointegration? A Prospective Multicenter Clinical Study Using Intraoral Scan Superimposition and Stability Analysis.
Brief Title: Movement of Dental Implants During Osseointegration
Acronym: MOVs-OI
Status: Not yet recruiting | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, PhD, Aula Dental Avanzada
Other Study IDs: MOVSOI
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dental Implants; Osseointegration
Keywords: Dental implants; Osseointegration; Intraoral scan; Micromotion; ISQ; Insertion torque; Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults receiving a single dental implant: Consecutive adults indicated for a single implant-supported restoration treated in three private clinics in Spain. Care follows standard practice; no investigational interventions are mandated. The exposure of interest is the osseointegration period between implant placement (T0) and pre-loading (T1, ~3-4 months). At T0 and T1, intraoral scans (STL) are acquired and rigidly superimposed with certified software to quantify 3D positional change (linear, mm; angular, degrees). Clinical variables recorded include insertion torque, ISQ1/ISQ2, anatomical site (jaw/region), placement timing (immediate/delayed), operator-perceived bone density, and bruxism/night-guard use. Analyses are performed at the implant level (one implant per participant).

SUMMARY:
Prospective multicenter observational study assessing whether dental implants undergo three-dimensional positional change between placement (T0) and pre-loading after osseointegration (T1). Two intraoral scans (STL) will be superimposed to quantify linear (mm) and angular (degrees) displacement. Clinical variables include insertion torque, primary and secondary ISQ, anatomical site, placement timing, operator-perceived bone density (Lekholm & Zarb), bruxism, and night guard use. The primary endpoint is the 3D displacement at ~3-4 months. Multivariable analyses will explore associated factors.

DETAILED DESCRIPTION:
This is a prospective multicenter observational study designed to evaluate whether dental implants undergo measurable three-dimensional positional changes during the osseointegration period. The study will be conducted in three private dental clinics in Spain, each led by an experienced implantologist. Consecutive adult patients indicated for a single implant-supported restoration will be enrolled after providing written informed consent.

Immediately after implant placement (T0), a reference intraoral scan (STL format) will be obtained using a validated scanner. A second intraoral scan will be performed after approximately 3 to 4 months, prior to prosthetic loading (T1). The two STL datasets will be superimposed using certified metrology software to calculate both linear (mm) and angular (degrees) displacement of the implant position relative to stable reference structures. The software alignment protocol ensures a reproducible and rigid registration of both scans.

Clinical and procedural variables collected at surgery include insertion torque value (ITV), primary implant stability (ISQ1), implant site (maxilla or mandible; anterior, premolar, or molar region), timing of placement (immediate or delayed), and operator-perceived bone density according to the Lekholm and Zarb classification. At the pre-loading visit (T1), secondary stability (ISQ2) will be recorded together with information on bruxism and the use of night guards.

The primary outcome is the 3D positional change (linear and angular) of the implant between T0 and T1. Secondary outcomes include the evolution of implant stability (ISQ2-ISQ1), correlations between displacement and insertion torque, and the influence of anatomical and patient-related variables (site, bone quality, bruxism, and loading protocol) on implant micromotion.

All data will be anonymized and analyzed at the implant level. Descriptive statistics will summarize means, standard deviations, and confidence intervals. Paired comparisons will be used to test within-subject changes, and multivariable linear regression models will explore predictors of displacement. Statistical significance will be set at p < 0.05.

The results of this study are expected to contribute to understanding whether clinically relevant implant micromovement occurs during osseointegration and to identify factors influencing this phenomenon, potentially guiding decisions on early loading and implant design optimization.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Indication for a single implant-supported restoration.
* Good general health and absence of active periodontal disease.
* Willingness to provide written informed consent and to undergo two intraoral scans (immediately after implant placement - T0 - and before prosthetic loading - T1).

Exclusion Criteria:

* Uncontrolled systemic disease or any medical condition contraindicating implant surgery.
* High-risk antiresorptive therapy (e.g., intravenous bisphosphonates or denosumab).
* Pregnancy or breastfeeding, if applicable to local policy.
* Inability to attend the T1 follow-up visit or contraindication to intraoral scanning (e.g., limited mouth opening, severe gag reflex).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients in good general health who require a single dental implant-supported restoration in private clinical practice. Participants will be recruited from three collaborating dental clinics in Spain (Alicante, Murcia, and Tenerife). All candidates will be screened according to inclusion and exclusion criteria and will receive standard implant therapy under routine clinical conditions. Each participant contributes one implant, which constitutes the analytical unit of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
3D positional change (linear and angular) from T0 to T1 | 3-4 months post-placement (pre-loading visit).
  Linear displacement (mm) and angular change (degrees) assessed by superimposing post-surgical (T0) and pre-loading (T1) intraoral STL scans using certified software.

SECONDARY OUTCOMES:
Change in implant stability (ISQ2 vs. ISQ1) | 3-4 months after implant placement (pre-loading visit).
  Difference in implant stability values measured by resonance frequency analysis between placement (ISQ1) and pre-loading (ISQ2). The mean ISQ gain will be analyzed and correlated with the magnitude of 3D displacement.
Association between 3D displacement and insertion torque | 3-4 months after implant placement.
  Evaluation of the correlation between linear and angular displacement (T0-T1) and the insertion torque value (ITV) recorded at implant placement. The aim is to determine whether higher primary mechanical stability predicts lower micromotion during osseointegration.
Proportion of implants with linear displacement >0.15 mm | 3-4 months after implant placement.
  Percentage of implants showing a linear displacement greater than 0.15 mm between T0 and T1, considered an exploratory biological threshold of potential micromotion. Sensitivity analyses will also be conducted using alternative thresholds (0.10-0.20 mm).
Influence of anatomical, surgical, and patient-related variables on 3D displacement | 3-4 months after implant placement.
  Multivariable analysis evaluating the influence of anatomical site (maxilla/mandible; anterior/premolar/molar), timing of placement (immediate/delayed), operator-perceived bone density (Lekholm & Zarb), and bruxism/night-guard use on 3D implant displacement.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Clínica Dental Esteve, Alicante, Alicante
  - Clínica Dental Sánchez Nicolás, Cabezo de Torres, Murcia
  - Clínica Dental García Marí, Santa Cruz de Tenerife, Tenerife

IPD SHARING:
Plan to Share IPD: Yes
De-identified implant-level and patient-level data will be made available upon reasonable request after publication of the main study results. Shared materials will include the full dataset (excluding any directly identifying information), the data dictionary, and the main statistical analysis code. Access requests must be submitted in writing to the study sponsor (Clínica Dental Esteve, S.L.) and will be reviewed by the principal investigator to ensure compliance with ethical and privacy regulations. Data will be provided through a secure repository or encrypted transfer.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning 6 months after publication of the primary results and for a minimum of 5 years thereafter.
Access Criteria: Qualified researchers affiliated with academic or non-profit institutions may request access to de-identified implant-level and patient-level data, the data dictionary, and the main analysis code. Requests must include a brief research proposal and be submitted in writing to the study sponsor (Clínica Dental Esteve, S.L.). The principal investigator will review each request for scientific merit and ethical compliance. Approved users will sign a data use agreement and receive secure, time-limited access through an encrypted repository managed by the sponsor.